CLINICAL TRIAL: NCT06869785
Title: An Open-label, Randomized, Parallel Group, Non-inferiority Study to Investigate the Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of a New Maintenance Dosing Regimen of Ofatumumab, Followed by Extended Treatment in Participants With Relapsing Multiple Sclerosis
Brief Title: Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of a New Maintenance Dosing Regimen of Ofatumumab
Acronym: FILIOS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COMB157Q12301
Record Dates: First submitted 2025-03-10; First posted 2025-03-11 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Relapsing Multiple Sclerosis (RMS)
Keywords: Relapsing Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ofatumumab dose 1 (Active Comparator): Approved dosage
  Interventions: Biological: Ofatumumab approved dose; Biological: Ofatumumab new dose
- Ofatumumab dose 2 (Experimental): New dosage
  Interventions: Biological: Ofatumumab new dose

INTERVENTIONS:
Biological: Ofatumumab approved dose — Approved dosage
  Arms: Ofatumumab dose 1
Biological: Ofatumumab new dose — New dosage

SUMMARY:
This study will evaluate the pharmacokinetics, pharmacodynamics, safety and tolerability of a new dosage of ofatumumab compared to the approved dosage of ofatumumab followed by extended treatment in participants with relapsing multiple sclerosis.

DETAILED DESCRIPTION:
This is a Phase 3, open label, parallel-group, multicenter study in participants with relapsing multiple sclerosis

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study.
* Male or female study participants aged 18 to 60 years (inclusive) at screening.
* Diagnosis of multiple sclerosis (MS) according to the 2017 Revised McDonald criteria (Thompson et al 2018). Relapsing forms of MS: relapsing-remitting MS (RRMS), or active secondary progressive MS (SPMS).

Exclusion Criteria:

* Participants suspected of not being able or willing to cooperate or comply with study protocol requirements in the opinion of the Investigator or emergence of any clinically significant condition/disease (e.g. active systemic bacterial, viral or fungal infections) during screening prior to Day 1 which might result in safety risk for participants.
* Participants with history of confirmed progressive multifocal leukoencephalopathy (PML) or neurological symptoms consistent with PML.
* Participants at risk of developing or having reactivation of hepatitis
* Emergence of active chronic disease (or stable but treated with immune therapy) prior to Day 1 of the immune system other than MS (e.g. rheumatoid arthritis, scleroderma, Sjögren's syndrome, Crohn's disease, ulcerative colitis, etc.) or with immunodeficiency syndrome (hereditary immune deficiency, drug-induced immune deficiency).
* Pregnant or nursing (lactating) women
* History of lymphoproliferative disease or any known malignancy or history of malignancy of any organ system (except for basal cell carcinoma, or squamous cell carcinomas of the skin that have been treated with no evidence of recurrence in the past 3 months).
* Participants taking prohibited therapies, including B cell targeted therapies (e.g. such as ocrelizumab, rituximab, ofatumumab, ublituximab, and inebilizumab)

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2026-12-24 (Estimated); Study Completion 2031-05-26 (Estimated)

PRIMARY OUTCOMES:
Ofatumumab plasma pharmacokinetics - area under the curve | Up to 12 weeks

SECONDARY OUTCOMES:
Ofatumumab plasma pharmacokinetics - minimum observed plasma concentration | Up to 12 weeks
Ofatumumab plasma pharmacokinetics - maximum observed plasma concentration | Up to 12 weeks
Incidence of Adverse events (AE) and Serious adverse events (SAE) | Up to 52 weeks
Proportion of participants with anti-drug antibodies | Up to 52 weeks
Participant B cell counts | Up to 52 weeks

CONTACTS AND LOCATIONS:
Locations (80):
- United States (78):
  - Alabama Neurology Associates PC, Birmingham, Alabama
  - Gilbert Neurology, Gilbert, Arizona
  - Xenoscience Inc, Phoenix, Arizona
  - Ctr for Neurology and Spine, Phoenix, Arizona
  - Phoenix Neurological Associates, Phoenix, Arizona
  - The Research and Education Inst. of Alta Bates Summit Med. Grp, Berkeley, California
  - Fullerton Neuro and Headache Ctr, Fullerton, California
  - University of California Irvine, Irvine, California
  - CenExcel Clinical Research, Los Alamitos, California
  - Velocity Clinical Trials, Los Angeles, California
  - Amicis Research Center, Valencia, California
  - Regina Berkovich MD PhD Inc, West Hollywood, California
  - CU Anschutz Med Campus, Aurora, Colorado
  - Mountain Neuro Research Center PC, Basalt, Colorado
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Neurology of Central FL Res Ctr, Altamonte Springs, Florida
  - Neurology Offices Of South Florida, Boca Raton, Florida
  - Baptist Health South Florida, Boca Raton, Florida
  - First Choice Neurology, Boca Raton, Florida
  - University of Florida, Gainesville, Florida
  - Memorial Healthcare System, Hollywood, Florida
  - Baptist Health Research Institute, Jacksonville, Florida
  - Neurology Associates PA, Maitland, Florida
  - UM Department Of Neurology, Miami, Florida
  - Elite Clinical Research, Miami, Florida
  - Reliant Medical Research, Miami, Florida
  - Aqualane Clinical Research, Naples, Florida
  - AdventHealth, Orlando, Florida
  - Orlando Health Clinical Trials, Orlando, Florida
  - Neurology Associates of Ormond Beach, Ormond Beach, Florida
  - Neurostudies Inc, Port Charlotte, Florida
  - Tallahassee Neurological Clinic, Tallahassee, Florida
  - Axiom Brain Health, Tampa, Florida
  - University Of South Florida, Tampa, Florida
  - Vero Beach Neurology, Vero Beach, Florida
  - Premiere Research Institute, West Palm Beach, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Atlanta NeuroScience Institute, Atlanta, Georgia
  - Insight Hospital and Medical Center, Chicago, Illinois
  - Josephson Wallack Munshower Neurology P.C, Indianapolis, Indiana
  - Univ of Kansas Hosp and Med Ctr, Kansas City, Kansas
  - Advent Neurology Clinic, Roeland Park, Kansas
  - Neuro Medial Clinic of Central Louisiana, Alexandria, Louisiana
  - Delricht Research, New Orleans, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - American Oncology Partners PA Center for Cancer & Blood Disorders, Bethesda, Maryland
  - International Neurorehab Institute, Lutherville, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - Trinity Health Michigan, Grand Rapids, Michigan
  - Rochester Cent For Behavioral, Rochester Hills, Michigan
  - WA Uni School Of Med, St Louis, Missouri
  - Cleveland Clinic Foundation, Las Vegas, Nevada
  - Hackensack University Medical Ctr, Hackensack, New Jersey
  - Jersey Shore University Medical Ctr, Neptune City, New Jersey
  - MS Comprehensive Care Ctr at Holy Name Hospi, Teaneck, New Jersey
  - Mount Sinai School Of Medicine, New York, New York
  - South Shore Neurologic Associates, Patchogue, New York
  - True North Neurology, Port Jefferson, New York
  - Atrium Health, Charlotte, North Carolina
  - Velocity Clinical Research, Raleigh, North Carolina
  - Dayton Center for Neurological Disorders, Centerville, Ohio
  - University Of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - OSU Medical Center-Martha Morehouse Medical Plaza, Columbus, Ohio
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Neurology Clinic PC, Cordova, Tennessee
  - University of Tennessee Medical Ctr, Knoxville, Tennessee
  - Sibyl Wray MD Neurology PC, Knoxville, Tennessee
  - Vanderbilt Comprehensive Multiple Sclerosis Center, Nashville, Tennessee
  - Texas Neurology, Dallas, Texas
  - Neurology Consultants Of Dallas PA, Dallas, Texas
  - Saturn Research Solutions LLC, Plano, Texas
  - Sana Research, Arlington, Virginia
  - Sentara Neuroscience Institute, Virginia Beach, Virginia
  - Swedish Neuroscience Institute, Seattle, Washington
  - MultiCare Research Institute for Research and Innovation, Tacoma, Washington
  - Gamma Therapeutic Center, Greenfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Puerto Rico (2):
  - Puerto Rico Multiple Sclerosis Ctr, Caguas
  - Caribbean Center for Clinical Research, Inc, Guaynabo

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.